CLINICAL TRIAL: NCT06964438
Title: A Three-Arm Randomised Controlled Trial to Establish Effectiveness of NMES With or Without Protein Supplementation to Preserve Muscle Mass and Strength and Improve Functional Outcomes After Abdominal Surgery for GI Cancer
Brief Title: Postoperative Electrical Muscle Stimulation Two
Acronym: POEMS2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24058; 347923 (Other: IRAS)
Record Dates: First submitted 2025-04-22; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Surgery; Colorectal Cancer; Muscle Atrophy; Cancer Gi
Keywords: electrical stimulation; neuromuscular electrical stimulation; NMES; rehabilitation; general surgery; colorectal surgery; laparotomy; laparoscopy; postoperative recovery; gastrointestinal cancer; gastrointestinal surgery
MeSH Terms: conditions — Colorectal Neoplasms; Muscular Atrophy; Gastrointestinal Neoplasms | interventions — Electric Stimulation

STUDY DESIGN:
Masking Description: Researchers running the trial and interacting with participant will not be blinded.
  Participant will be blinded regarding protein drink allocation but not regarding NMES allocation.
  The assessor of the primary outcome (ultrasound VL measurements) will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 - Control (No Intervention): Standard postoperative care days 1-4
- Group 2 - NMES (no protein drink) (Experimental): Standard postoperative care days 1-4 PLUS twice daily NMES training sessions PLUS placebo drink twice daily (no protein supplement)
  Interventions: Device: Neuromuscular Electrical Stimulation
- Group 3 - NMES + protein drink (Experimental): Standard postoperative care days 1-4 PLUS twice daily NMES training sessions PLUS protein drink twice daily
  Interventions: Device: Neuromuscular Electrical Stimulation; Dietary Supplement: Protein supplement drink

INTERVENTIONS:
Device: Neuromuscular Electrical Stimulation — Neuromuscular Electrical Stimulation training twice daily (30 minutes per session), during postoperative days 1-4. The training will be carried out using a handheld device. Training will be carried out by the participant themselves, with researcher supervision until independently able to do so.
  Other Names: NMES; electrical stimulation; ES; electrical muscle stimulation; EMS
  Arms: Group 2 - NMES (no protein drink); Group 3 - NMES + protein drink
Dietary Supplement: Protein supplement drink — Whey protein isolate drink, to provide a total of 60 g protein per day (2 x30 g).
  The supplement will be provided in a powder form to participants. Participants will be asked to consume the supplement around the time of NMES training.
  Arms: Group 3 - NMES + protein drink

SUMMARY:
Undesirable loss of skeletal muscle mass (atrophy) is a common feature of many diseases as well as ageing, bed rest and physical inactivity. Losing muscle can lead to a reduction in one's ability to perform physical activities, and reduce independence and overall health. Muscle mass loss occurs very quickly (i.e., within a few days) after surgery.

The investigators previous work has shown that neuromuscular electrical stimulation (NMES) of the thigh muscles on one side of the body can help maintain muscle mass and strength on the stimulated side after surgery. Since then, additional work has been carried out to find the most effective form of stimulation to build muscle.

The current study aims to use this refined stimulation protocol in a clinical trial on the wards after major abdominal surgery. The intervention will involve delivering stimulation to both thighs in the few days after surgery, so that the investigators can assess whether this stimulation can preserve muscle mass and strength, and also, patients' ability to perform physical activities after surgery. In addition, the study will aim to find out whether any benefit provided by electrical stimulation can be increased further by taking a protein supplement at the same time.

DETAILED DESCRIPTION:
The main objective of this trial is to assess whether neuromuscular stimulation (NMES) can minimise muscle loss following abdominal surgery for cancer; and whether such effect is further improved by simultaneous protein supplementation.

The main questions it aims to answer are:

* Does NMES training reduce the volume of muscle lost from the vastus lateralis (VL) muscle (in the thigh) after surgery as measured on ultrasound scan 5 days after surgery?
* Does NMES training together with protein supplementation lead to greater reduction of VL muscle volume loss on ultrasound 5 days after surgery then NMES alone?

Researchers will allocate participants into three groups (using a randomisation software).

All participants will visit the hospital once before surgery for starting point measurements including ultrasound.

Whilst they are in hospital, from the first until the fourth day after surgery, they will have the following interventions:

* Group 1 (the control group) will receive usual post-operative care with no additional interventions;
* Group 2 will receive normal postoperative care and twice daily NMES training sessions and a flavoured (placebo) drink
* Group 3 will receive normal post operative care as well as twice daily NMES training sessions and two protein rich drinks per day.

On the fifth day after surgery all participants will have repeat measurements including ultrasound to assess the extent of muscle loss they had since surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 or over at the time of diagnosis made at MDT (multi-disciplinary team meeting)
* MDT outcome of colorectal or gastric cancer or non-invasive neoplasia (tissue-proven, or radiologically diagnosed and clinically suspected) with the intention to treat with curative abdominal surgery
* Agreed management plan for open or minimally invasive (laparoscopic or robot assisted) segmental abdominal (colonic or gastric) resection at the Royal Derby Hospital
* Sufficient mobility and fitness to complete normal ERAS (enhanced recovery after surgery) protocols following surgery
* Basic conversational spoken English language
* Ability to give informed consent

Exclusion Criteria:

* Upper GI (gastrointestinal) cancer requiring thoracotomy/thoracoscopy
* Pre-existing neuromuscular disease (including Parkinsons disease)
* Pacemaker, implantable cardiac defibrillator or other implanted nerve stimulator device
* Metal prostheses or other metal-work in either upper legs (hip/knee/femur)
* Dementia or other cognitive problem or language barrier causing an inability to follow instructions and operate NMES machine
* Inability to give informed consent
* Disability preventing completion of ERAS after surgery (requiring Zimmer frame/wheeled frame/wheelchair to mobilise or bed-bound)
* Peripheral vascular disease
* Epilepsy
* Pre-existing diagnosis of chronic kidney disease or estimated glomerular filtration rate <60 on screening visit
* Pre-existing diagnosis of liver disease
* Intubation or intensive care admission during study period (between day 0-5 post-op); (surgical high dependency unit patients will be included)
* Return to theatre for surgical complication within first 5-days post operation
* History of rhabdomyolysis
* Pregnancy
* Deep vein thrombosis within past 6-months
* Allergy to whey protein
* Patient refusal of whey protein products on grounds of dietary requirements or intolerance
* Participating in another clinical trial concurrently or within the last 6 months
* Known infection with blood borne virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Post-operative vastus lateralis (VL) muscle mass loss | Pre-operatively and 5 days post-operatively
  Vastus lateralis (VL) muscle mass loss as measured on ultrasound cross sectional area

SECONDARY OUTCOMES:
Post-operative knee extensor strength losses | Pre-operatively and 5 days post-operatively
  Determined by knee-extensor strength via dynamometry.
Post-operative functional losses determined by short physical performance battery standardized physical function assessment tool | Pre-operatively and 5 days post-operatively
  short physical performance battery
Post-operative functional losses determined by Timed Up and Go standardized physical function assessment tool | Pre-operatively and 5 days post-operatively
  Timed up and go,
Post-operative functional losses determined by 6 minute walk test standardized physical function assessment tool | Pre-operatively and 5 days post-operatively
  6 minute walk test
Post-operative changes in muscle architecture as measured by pennation angle | Pre-operatively and 5 days post-operatively
  Pennation angle on VL US
Post-operative changes in muscle architecture as measured by fascicle length | Pre-operatively and 5 days post-operatively
  fascicle length on VL Ultrasound
Post-operative declines in neuromuscular function | Pre-operatively and 5 days post-operatively
  Determined via surface electromyography
Post-operative loss of independence and quality of life | Pre-operatively, 5 days post-operatively and 28 days post-operatively
  Measured using the EuroQoL-5D questionnaire. The EuroQoL-5D-3L questionnaire is a standardised measure of health status developed by the EuroQol Group to provide a simple, generic measure of health for clinical and economic appraisal. It generates a simple descriptive profile and a single summary index value for health status.
Physical activity profiles of patients following major GI surgery | Days 1-4 post operatively
  Measured using a thigh-worn accelerometer
Circulating amino acid profiles | Pre-operatively, and on day 1 and 5 post-operatively
  Blood samples to assess circulatory amino acid levels
Systemic markers of inflammation | Pre-operatively, and on day 1 and 5 post-operatively
  Blood samples to assess inflammatory marker levels
Post-operative vastus lateralis (VL) muscle mass loss | Pre-operatively and 5 days post-operatively
  Vastus lateralis (VL) muscle mass loss as measured on ultrasound muscle thickness

OTHER OUTCOMES:
Feasibility and acceptability of incorporating NMES into postoperative recovery | Days 1-4 post-operatively
  Assessed through compliance and participant feedback questionnaire. The questionnaire will compromise descriptive items rated on a visual analogue scale that has been designed by the researchers to assess various aspects of patient experience with the intervention.

IPD SHARING:
Plan to Share IPD: No